CLINICAL TRIAL: NCT05969314
Title: Phase I Study of Safety and Feasibility of Ayurvedic Oral Cannabis Preparation in the Peri-operative Period in Breast and Oral Cavity Squamous Cell Cancer
Brief Title: To Check Safety of Ayurvedic Oral Cannabis in Breast and Head and Neck Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Dr Rajendra A. Badwe, Doctor, Tata Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMH Project No. 3386; CTRI/2020/06/020649 (Registry Identifier: Clinical Trials Registry of India)
Record Dates: First submitted 2022-05-31; First posted 2023-08-01 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer; Oral Cancer
MeSH Terms: conditions — Breast Neoplasms; Mouth Neoplasms | interventions — nabiximols

STUDY DESIGN:
Intervention Model Description: To determine the maximum tolerated dose (MTD). First 3 patients will receive the study preparation once a day at 9 am (+/- 60 min) (i.e 5 mg of CBD and 5 mg of THC in a 400 mg capsule). Subsequent cohorts will be administered doses of 10 (10 mg of THC and CBD each), 20 (20+20) and 30 (30+30) mg in a classical 3+3 dose escalation study. Briefly, 3 patients will be enrolled at dose level. Dose escalation to the next dose level will continue as long no DLT is observed in 3 patients (the incidence of DLT is ≤ 1/6) In any cohort, if 1/3 patients develop DLT, then 3 more patients will be added at that dose. The dose level at which more than 1/6 patients develop DLT will be considered the MTD and no further escalation will be done beyond the MTD. One dose level below the MTD will be considered for future trials. If MTD is not achieved, the highest dose (30+30) will be considered for future trials. If toxicity is seen at 30 mg, then de-escalation to 25 mg may be considered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cannabis (Experimental): Cannabis capsules containing 5 mg of THC and CBD each or 2.5 mg of THC and CBD each.
  Interventions: Drug: Cannabis capsules

INTERVENTIONS:
Drug: Cannabis capsules — Cannabis capsules containing 5 mg of THC and CBD each or 2.5 mg of THC and CBD each.

SUMMARY:
Phase 1 study to assess the pharmacokinetic availability and safety and tolerability profile of one such ayurvedic preparation which contains 5 mg THC:CBD 1:1 preparation. Other than the PK profile, we will also be studying its effect on gene expression profiling of the breast and head neck oral cavity squamous cell carcinoma tissue.

DETAILED DESCRIPTION:
The ancient Ayurvedic medicine obtained from Cannabis sativa plant has recently been re-explored for its anti-inflammatory and anti-cancer potential. Various laboratory and preclinical studies have proven its anti-cancer activity and its effect on all the hallmarks of cancer. Anecdotal clinical evidence has shown regression of tumours with ingestion of such medicinal cannabis. A randomized controlled trial in Glioblastoma Multiforme, a kind of brain tumour, shows improvement in disease free survival when temozolamide was combined with Cannabis spray called Sativex.

However, because of lack of systematic, large volume studies, the evidence is slow to emerge. We have previously seen changes related to NF-kb (inflammation) and AP1 (acute hypoxia/stress) pathway genes within the tumour tissue as assessed by transcriptomic analysis (Yet unpublished data). There is laboratory evidence to suggest that the changes induced in the AP1 pathway during surgery can be ameliorated by cannabis treatment. We intend to explore this anticancer potential of C sativa herbal preparation in the pre-operative setting in breast and head and neck cancer patients. Hence, we are proposing a phase 1 study to assess the pharmacokinetic availability and safety and tolerability profile of one such ayurvedic preparation which contains 5 mg THC:CBD 1:1 preparation. Other than the PK profile, we will also be studying its effect on gene expression profiling of the breast and head neck oral cavity squamous cell carcinoma tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically proven patients of breast or oral cavity SCC
2. Age > 18 and < 65
3. Operable cancers planned to undergo upfront curative surgery
4. Patient fit for surgery (ASA Grade I / II)
5. Patient Voluntarily willing to give consent for study

Exclusion Criteria:

1. Planned for any other pre or peri-operative intervention such as neoadjuvant chemotherapy or targeted therapy or radiation
2. Presence of medical disease such as pulmonary, renal, liver, gastro-intestinal disease which may interfere with any study specific procedure (deranged renal parameters > 1.5 times normal range or deranged liver function tests such as > 2.5 times raised liver enzymes)
3. History of substance abuse (including cannabis-related products) or alcohol abuse
4. Personal history of psychiatric disease or Significant family history of psychiatric disease
5. Pregnancy and/or lactation
6. Patients currently (within last 14 days before consenting) on other CNS depressants such as alcohol, barbiturates, benozodiazapines (like diazepam, alprazolam etc)
7. Patients on other medications which will likely have a drug interaction with cannabis- such as clozapine, duloxetine, naproxen, cyclobenzaprine, olanzapine, haloperidol, and chlorpromazine, macrolides, calcium channel blockers, benzodiazepines, cyclosporine, sildenafil (and other PDE5 inhibitors), antihistamines, haloperidol, antiretrovirals
8. Any other illness or abnormal laboratory investigations which the investigator considers as making the patients ineligible for the study
9. Any patient with positive HIV, HBsAg, HCV status

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
To establish safe dose of oral cannabis preparation | From day 1 of IP dosing till 28 days .
  Number of participants with treatment-related adverse events with respect to cardiovascular, central nervous system and psychotropic of cannabis as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Pharmacokinetic profiling | 1.Pre operative day 1 to 5 - one each day before cannabinoid dosing, after dosing 30 minutes, 1 hour, 2 hour and 8 hour. 2. On day of surgery - Before and after the surgery 3. Post operative day 1 , day 2, day 3 and day 14
  Blood samples collected during the administration of the IP for 5 days and up to 72 hours after surgery.
Biomarker analysis- Transcitpomics | A baseline pre-cannabis tumor tissue sample will be collected before starting IP(day 0). Further blood and tumor as well as adjacent normal tissue samples will be collected during surgery (day6).
  Tumor and normal tissue samples.

CONTACTS AND LOCATIONS:
Overall Officials: Rajendra A Badwe, MS, Principal Investigator — Director, Tata Memorial Centre
Locations (2):
- India (2):
  - Tata Memorial Center, Mumbai, Maharashtra
  - Tata Memorial Hospital, Mumbai, Maharashtra

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zuardi AW. History of cannabis as a medicine: a review. Braz J Psychiatry. 2006 Jun;28(2):153-7. doi: 10.1590/s1516-44462006000200015. Epub 2006 Jun 26. PMID 16810401
- [Background] ElSohly MA, Radwan MM, Gul W, Chandra S, Galal A. Phytochemistry of Cannabis sativa L. Prog Chem Org Nat Prod. 2017;103:1-36. doi: 10.1007/978-3-319-45541-9_1. PMID 28120229
- [Background] Ben Amar M. Cannabinoids in medicine: A review of their therapeutic potential. J Ethnopharmacol. 2006 Apr 21;105(1-2):1-25. doi: 10.1016/j.jep.2006.02.001. Epub 2006 Mar 15. PMID 16540272
- [Background] Whiting PF, Wolff RF, Deshpande S, Di Nisio M, Duffy S, Hernandez AV, Keurentjes JC, Lang S, Misso K, Ryder S, Schmidlkofer S, Westwood M, Kleijnen J. Cannabinoids for Medical Use: A Systematic Review and Meta-analysis. JAMA. 2015 Jun 23-30;313(24):2456-73. doi: 10.1001/jama.2015.6358. PMID 26103030
- [Background] Bar-Sela G, Vorobeichik M, Drawsheh S, Omer A, Goldberg V, Muller E. The medical necessity for medicinal cannabis: prospective, observational study evaluating the treatment in cancer patients on supportive or palliative care. Evid Based Complement Alternat Med. 2013;2013:510392. doi: 10.1155/2013/510392. Epub 2013 Jul 16. PMID 23956774
- [Background] Waissengrin B, Urban D, Leshem Y, Garty M, Wolf I. Patterns of use of medical cannabis among Israeli cancer patients: a single institution experience. J Pain Symptom Manage. 2015 Feb;49(2):223-30. doi: 10.1016/j.jpainsymman.2014.05.018. Epub 2014 Jun 14. PMID 24937161
- [Background] Vara D, Salazar M, Olea-Herrero N, Guzman M, Velasco G, Diaz-Laviada I. Anti-tumoral action of cannabinoids on hepatocellular carcinoma: role of AMPK-dependent activation of autophagy. Cell Death Differ. 2011 Jul;18(7):1099-111. doi: 10.1038/cdd.2011.32. Epub 2011 Apr 8. PMID 21475304
- [Background] Caffarel MM, Sarrio D, Palacios J, Guzman M, Sanchez C. Delta9-tetrahydrocannabinol inhibits cell cycle progression in human breast cancer cells through Cdc2 regulation. Cancer Res. 2006 Jul 1;66(13):6615-21. doi: 10.1158/0008-5472.CAN-05-4566. PMID 16818634
- [Background] Caffarel MM, Moreno-Bueno G, Cerutti C, Palacios J, Guzman M, Mechta-Grigoriou F, Sanchez C. JunD is involved in the antiproliferative effect of Delta9-tetrahydrocannabinol on human breast cancer cells. Oncogene. 2008 Aug 28;27(37):5033-44. doi: 10.1038/onc.2008.145. Epub 2008 May 5. PMID 18454173
- [Background] Salazar M, Carracedo A, Salanueva IJ, Hernandez-Tiedra S, Lorente M, Egia A, Vazquez P, Blazquez C, Torres S, Garcia S, Nowak J, Fimia GM, Piacentini M, Cecconi F, Pandolfi PP, Gonzalez-Feria L, Iovanna JL, Guzman M, Boya P, Velasco G. Cannabinoid action induces autophagy-mediated cell death through stimulation of ER stress in human glioma cells. J Clin Invest. 2009 May;119(5):1359-72. doi: 10.1172/jci37948. PMID 19425170
- [Background] Lopes CF, de Angelis BB, Prudente HM, de Souza BV, Cardoso SV, de Azambuja Ribeiro RI. Concomitant consumption of marijuana, alcohol and tobacco in oral squamous cell carcinoma development and progression: recent advances and challenges. Arch Oral Biol. 2012 Aug;57(8):1026-33. doi: 10.1016/j.archoralbio.2012.05.006. Epub 2012 Jun 22. PMID 22727410
- [Background] Cozzolino R, Cali G, Bifulco M, Laccetti P. A metabolically stable analogue of anandamide, Met-F-AEA, inhibits human thyroid carcinoma cell lines by activation of apoptosis. Invest New Drugs. 2010 Apr;28(2):115-23. doi: 10.1007/s10637-009-9221-0. Epub 2009 Feb 3. PMID 19189054
- [Background] Badwe R, Hawaldar R, Parmar V, Nadkarni M, Shet T, Desai S, Gupta S, Jalali R, Vanmali V, Dikshit R, Mittra I. Single-injection depot progesterone before surgery and survival in women with operable breast cancer: a randomized controlled trial. J Clin Oncol. 2011 Jul 20;29(21):2845-51. doi: 10.1200/JCO.2010.33.0738. Epub 2011 Jun 13. PMID 21670457
- [Background] Chakravarti B, Ravi J, Ganju RK. Cannabinoids as therapeutic agents in cancer: current status and future implications. Oncotarget. 2014 Aug 15;5(15):5852-72. doi: 10.18632/oncotarget.2233. PMID 25115386
- [Background] Nagarkatti P, Pandey R, Rieder SA, Hegde VL, Nagarkatti M. Cannabinoids as novel anti-inflammatory drugs. Future Med Chem. 2009 Oct;1(7):1333-49. doi: 10.4155/fmc.09.93. PMID 20191092
- [Background] Ohlsson A, Lindgren JE, Wahlen A, Agurell S, Hollister LE, Gillespie HK. Plasma delta-9 tetrahydrocannabinol concentrations and clinical effects after oral and intravenous administration and smoking. Clin Pharmacol Ther. 1980 Sep;28(3):409-16. doi: 10.1038/clpt.1980.181. PMID 6250760
- [Background] Karschner EL, Darwin WD, Goodwin RS, Wright S, Huestis MA. Plasma cannabinoid pharmacokinetics following controlled oral delta9-tetrahydrocannabinol and oromucosal cannabis extract administration. Clin Chem. 2011 Jan;57(1):66-75. doi: 10.1373/clinchem.2010.152439. Epub 2010 Nov 15. PMID 21078841
- [Background] Atsmon J, Heffetz D, Deutsch L, Deutsch F, Sacks H. Single-Dose Pharmacokinetics of Oral Cannabidiol Following Administration of PTL101: A New Formulation Based on Gelatin Matrix Pellets Technology. Clin Pharmacol Drug Dev. 2018 Sep;7(7):751-758. doi: 10.1002/cpdd.408. Epub 2017 Nov 10. PMID 29125702
- [Background] Cherniakov I, Izgelov D, Domb AJ, Hoffman A. The effect of Pro NanoLipospheres (PNL) formulation containing natural absorption enhancers on the oral bioavailability of delta-9-tetrahydrocannabinol (THC) and cannabidiol (CBD) in a rat model. Eur J Pharm Sci. 2017 Nov 15;109:21-30. doi: 10.1016/j.ejps.2017.07.003. Epub 2017 Jul 20. PMID 28736128
- [Background] Manini AF, Yiannoulos G, Bergamaschi MM, Hernandez S, Olmedo R, Barnes AJ, Winkel G, Sinha R, Jutras-Aswad D, Huestis MA, Hurd YL. Safety and pharmacokinetics of oral cannabidiol when administered concomitantly with intravenous fentanyl in humans. J Addict Med. 2015 May-Jun;9(3):204-10. doi: 10.1097/ADM.0000000000000118. PMID 25748562
- [Background] Vandrey R, Herrmann ES, Mitchell JM, Bigelow GE, Flegel R, LoDico C, Cone EJ. Pharmacokinetic Profile of Oral Cannabis in Humans: Blood and Oral Fluid Disposition and Relation to Pharmacodynamic Outcomes. J Anal Toxicol. 2017 Mar 1;41(2):83-99. doi: 10.1093/jat/bkx012. PMID 28158482
- [Background] Bergamaschi MM, Queiroz RH, Zuardi AW, Crippa JA. Safety and side effects of cannabidiol, a Cannabis sativa constituent. Curr Drug Saf. 2011 Sep 1;6(4):237-49. doi: 10.2174/157488611798280924. PMID 22129319
- [Background] Zuardi AW, Shirakawa I, Finkelfarb E, Karniol IG. Action of cannabidiol on the anxiety and other effects produced by delta 9-THC in normal subjects. Psychopharmacology (Berl). 1982;76(3):245-50. doi: 10.1007/BF00432554. PMID 6285406
- [Background] Crippa JA, Zuardi AW, Garrido GE, Wichert-Ana L, Guarnieri R, Ferrari L, Azevedo-Marques PM, Hallak JE, McGuire PK, Filho Busatto G. Effects of cannabidiol (CBD) on regional cerebral blood flow. Neuropsychopharmacology. 2004 Feb;29(2):417-26. doi: 10.1038/sj.npp.1300340. PMID 14583744
- [Background] Fusar-Poli P, Crippa JA, Bhattacharyya S, Borgwardt SJ, Allen P, Martin-Santos R, Seal M, Surguladze SA, O'Carrol C, Atakan Z, Zuardi AW, McGuire PK. Distinct effects of delta9-tetrahydrocannabinol and cannabidiol on neural activation during emotional processing. Arch Gen Psychiatry. 2009 Jan;66(1):95-105. doi: 10.1001/archgenpsychiatry.2008.519. PMID 19124693
- [Background] Bhattacharyya S, Morrison PD, Fusar-Poli P, Martin-Santos R, Borgwardt S, Winton-Brown T, Nosarti C, O' Carroll CM, Seal M, Allen P, Mehta MA, Stone JM, Tunstall N, Giampietro V, Kapur S, Murray RM, Zuardi AW, Crippa JA, Atakan Z, McGuire PK. Opposite effects of delta-9-tetrahydrocannabinol and cannabidiol on human brain function and psychopathology. Neuropsychopharmacology. 2010 Feb;35(3):764-74. doi: 10.1038/npp.2009.184. Epub 2009 Nov 18. PMID 19924114
- [Background] Schubart CD, Sommer IE, van Gastel WA, Goetgebuer RL, Kahn RS, Boks MP. Cannabis with high cannabidiol content is associated with fewer psychotic experiences. Schizophr Res. 2011 Aug;130(1-3):216-21. doi: 10.1016/j.schres.2011.04.017. Epub 2011 May 17. PMID 21592732